CLINICAL TRIAL: NCT05892055
Title: Brain Mechanisms of Attention and Pain in Youth With Functional Abdominal Pain Disorders
Brief Title: Brain Mechanisms of Attention and Pain in Youth With FAPD
Status: Withdrawn | Type: Observational
Why Stopped: No participants were enrolled for the active phase of this study (with neuroimaging), but, n=6 (n=3 with FAPD and n=3 Healthy) completed the pilot testing protocol outside of the scanner between 2/28/2019 and 3/28/2019. No neuroimaging took place.
Sponsor: Michigan State University (Other)
Collaborators: Corewell Health West (Other)
Responsible Party: Principal Investigator, Natoshia Cunningham, Principal Investigator, Michigan State University
Other Study IDs: 2018-4315
Record Dates: First submitted 2019-02-19; First posted 2023-06-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Functional Abdominal Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control (HC): Healthy controls (HC) will not have an FAPD diagnosis. The HC group receives the same procedures as the FAPD group.
  Interventions: Other: MRI Procedure
- FAPD: Children in the FAPD group will be recruited based on the presence of an FAPD diagnosis and receive the same procedures as the HC group.
  Interventions: Other: MRI Procedure

INTERVENTIONS:
Other: MRI Procedure — All children will receive a functional magnetic resonance imaging (fMRI) scan, where they will complete some preliminary scans while completing two cognitive tasks, and then be removed from the scanner to complete a water loading symptom provocation task (WL-SPT). After the WL-SPT task, they will resume the fMRI scan and complete additional cognitive tasks to assess for diminished attentional regulation. Measures of pain intensity, pain unpleasantness, and state anxiety will be obtained throughout.

SUMMARY:
The objectives of this study are to identify neural mechanisms of increased pain in pediatric FAPD and examine mechanisms of disrupted attention in the presence of induced pain. The overarching goal is to determine whether youth with FAPD process pain differently than healthy youth and to identify the brain areas involved.

DETAILED DESCRIPTION:
The goal of the current project is to enhance understanding of the neural mechanisms associated with the pain experience in youth with functional abdominal pain disorders (FAPD), which is the most common and debilitating presentation of FAPD. This study will examine the neural mechanisms associated with pain induction and diminished attentional regulation during pain in FAPD. Findings from pilot studies indicate that increased anxiety in FAPD is associated with higher pain-related impairment, and that anxiety may adversely impact response to a cognitive behavioral intervention for pain. While pain outcomes improve when anxiety is also addressed in treatment for FAPD, a sizable portion fail to respond to currently available interventions. Further, the PI found that induced pain in FAPD is associated with changes in regional brain activity and functional connectivity between brain regions that are implicated in chronic pain. It is crucial to better understand the neural mechanisms which may place youth with FAPD at risk for poorer outcomes in order to ultimately develop more effective treatments. In this study, neural mechanisms of response to a pain symptom provocation task in youth with FAPD will be compared to healthy controls. The impact of anxiety levels will also be explored. This study will also examine neural mechanisms associated with disrupted attentional regulation during pain induction in youth with FAPD.

ELIGIBILITY:
Inclusion Criteria:

1. Children (boys and girls) between 11-16 years of age and their parent/primary caregiver.
2. Meets criteria for one of two study groups:

   * FAPD: based on physician diagnosis of FAPD confirmed by a validated Rome IV measure.
   * HC: based on a rule out of an FAPD diagnosis (using the Rome IV measure).

   We will recruit approximately 50% of HCs with and without clinical levels of anxiety (e.g,. SCARED cut-off score greater than or equal to 25) to match the anxiety levels anticipated in the FAPD group.
3. Sufficient English language ability necessary to complete study measures and protocol

Exclusion Criteria

1. Children with significant medical condition(s) with an identifiable organic cause including those that may account for abdominal pain symptoms (e.g., Inflammatory Bowel Diseases such as Ulcerative Colitis and Crohn's Disease). Rationale: Children with a significant medical condition may impact the study results. Further, youth with organic conditions that include abdominal pain may not meet criteria for FAPD even if they present with similar symptoms.
2. Children with a documented developmental delay, autism spectrum disorder, a previously diagnosed thought disorder (i.e., psychosis), or bipolar disorder will be excluded. Rationale: These comorbidities may confound the study aims by impacting the dependent measures.
3. Significant visual, hearing, or speech impairment. Rationale: Children will be excluded if they are not able to see the testing stimuli, hear the test examiner, or respond verbally to the test examiner, even with the help of corrective or assistive devices (e.g., glasses, hearing aids).
4. Organic brain injury. Rationale: Children must not have a history of epilepsy, a head trauma associated with a loss of consciousness, or any other organic disorder since these conditions could possibly affect brain function and cognition and interfere with study results.
5. *Other exclusionary criteria specific to the fMRI component of the study:

   * Participants with an implant such as a cochlear implant device, a pacemaker or neurostimulator containing electrical circuitry or generating magnetic signals will be excluded. Participants must also not have any significant ferrous material in their body that could pose the potential for harm in the fMRI environment or cause signal suppression of key regions (i.e. orthodontia). Rationale: Implant devices can malfunction and/or be damaged. Strong magnetic fields in the fMRI environment can cause some metallic objects to move and/or heat, and therefore pose a safety risk. All children will be screened prior to participation using a standardized questionnaire in the fMRI component of the study to ensure that the fMRI magnetic fields will not pose any risk to their safety.
   * Female participants who report current/suspected pregnancy will be excluded. Rationale: There is minimal yet potential fetal risk due to electromagnetic radiation from the MRI. Female participants who self-report that they may be pregnant will be excluded from the study.
   * Participants with evidence of claustrophobia will be excluded. Rationale: Such participants may experience extreme distress when entering the fMRI scanner. Claustrophobia will be assessed using a validated module of the Anxiety Disorders Interview Schedule as part of the initial screening process. Youth will be excluded from participating if they report excessive fear of enclosures.

     * Note that these exclusionary criteria do not apply to those recruited for the study's pilot portion.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 10 youth with be recruited to pilot test the procedures outside of the scanner (up to 5 HC and up to 5 with FAPD). Then, for the active part of the study, a total of 50 participants will be recruited (25 with FAPD and 25 HC). Children with FAPD will be recruited based on the presence of an FAPD diagnosis (see inclusion/exclusion criteria). Healthy controls (HC) will not have an FAPD diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Neural Mechanisms During Pain Induction | Approximately 1.5 hours
  Amygdala-Prefrontal Cortex (AMY-PFC) functional connectivity will be enhanced following WL-SPT in the FAPD group vs HC. Increased brain activity and functional connectivity will correspond to higher pain in FAPD.

SECONDARY OUTCOMES:
Attentional Regulation During Cognitive Task | Approximately 30 minutes
  Functional connectivity between the AMY-PFC will be enhanced during a cognitive task, which will be related to higher pain ratings and response time.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT05892055/Prot_SAP_000.pdf